CLINICAL TRIAL: NCT03758560
Title: Association of Preoperative Pain Catastrophizing With Postoperative Pain After Lower Limb Trauma Surgery
Brief Title: Preoperative Pain Catastrophizing and Its Association With Postoperative Pain After Lower Limb Trauma Surgery
Status: Completed | Type: Observational
Sponsor: B.P. Koirala Institute of Health Sciences (Other)
Responsible Party: Principal Investigator, Dr Asish Subedi, Principal Investigator, B.P. Koirala Institute of Health Sciences
Other Study IDs: IRC/1441/018
Record Dates: First submitted 2018-11-25; First posted 2018-11-29 (Actual); Last update posted 2019-09-09 (Actual); Status verified 2019-09

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Pre-operative Nepali version of pain catastrophizing scale (PCS) questionnaire — Patients will be asked to complete the scores based Nepali version of pain catastrophizing scale (PCS) questionnaire preoperatively

SUMMARY:
The Pain Catastrophizing Scale (PCS) is a psychometric tool to identify PC. A positive correlation between PCS scores and various pain outcomes has been reported in acute and chronic pain settings. Preoperative catastrophizing is associated with an increased intensity of postoperative pain and more analgesic consumption. Likewise, a recent meta-analysis revealed that PC is a strong predictor of persistent postsurgical pain. The Nepali version of PCS has been validated recently in patients with chronic pain. However, it has not been used in patients with acute pain. Therefore, our aim is to assess the relationship between preoperative Nepali PCS (N-PCS) scores and postoperative pain intensity and total opioid consumption in patients with musculoskeletal trauma planned for surgery.

DETAILED DESCRIPTION:
After approval from Institute Review Committee, we will assess eligibility of patients admitted in-patient-unit of orthopaedic ward planned for lower limb trauma surgery under spinal anesthesia. Recruited patients will be counseled and informed about the study and information sheet and consent form provided. Will obtain consent from the participant. patients will be asked to complete N- PCS questionnaire preoperatively a night before surgery in patient unit. On arrival to the operating room, standard monitoring will be applied. All the patients will receive spinal anaesthesia with 2.6 ml of hyperbaric bupivacaine (0.5%) and fentanyl 20 µg. NRS scale will be used to assess the intensity of their pain postoperatively on arrival to Post-anesthesia care unit, at 2, 4, 6, 12 h and 24 h after the end of surgery. One gram paracetamol IV and Ketorolac 30 mg IV will be given at the end of surgery and continued at 6 and 8 h intervals postoperatively. If the Numeric rating scale (NRS) for pain is > 3 at rest, tramadol 50 mg IV bolus administered, and repeated at 10 min intervals until NRS was ≤ 3 for the first 24 h. Patients will be asked to rate their worst or maximum pain intensity during the first 24 hours after surgery, on an 11-point numerical rating scale. Socio-demographic variables (age, BMI, ethnicity, gender, socio-economic status, occupation and education), preoperative anxiety of the participant will be recorded.

ELIGIBILITY:
Inclusion Criteria:

Patients with traumatic lower-limb injury scheduled for lower-extremity surgery under spinal anaesthesia.

American Society of Anaesthesiologists physical status I or II, Age between 18 and 65 years of age

Exclusion Criteria:

* Non- responders, Those unable to read and write; or Patients with known psychiatric disorder, Prior intake of pain medication, and Chronic pain.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with lower limb musculo-skeletal trauma admitted in the orthopaedic unit of BPKIHS and planned for elective surgery.
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2018-12-16 (Actual); Primary Completion 2019-08-16 (Actual); Study Completion 2019-09-03 (Actual)

PRIMARY OUTCOMES:
Correlation of preoperative pain catastrophizing scale (PCS) scores with maximum pain severity at 24 hrs post-operatively. | 24 hours postoperatively
  Correlation of preoperative pain catastrophizing scale scores with maximum pain severity at 24 hrs post-operatively. PCS consists of 13 items rated on a 5-point Likert scales from 0 (never) to 4 (all the time) points. The total score for the PCS is 52, with points more than 24 indicating a high level of catastrophizing. Worst or maximum pain intensity during the first 24 hours after surgery is assessed on an 11-point numerical rating scale (NRS). Pain is rated on a 0 to 11 NRS, with 0="no pain" or and 10=pain "as bad as you can imagine."

SECONDARY OUTCOMES:
Correlation between preoperative pain catastrophizing scale (PCS) scores with total tramadol consumption postoperatively at 24 hrs | 24 hrs postoperatively
  Correlation between preoperative pain catastrophizing scale scores with total tramadol consumption postoperatively upto 24 hrs. PCS consists of 13 items rated on a 5-point Likert scales from 0 (never) to 4 (all the time) points. The total score for the PCS is 52, with points more than 24 indicating a high level of catastrophizing.
Correlation of preoperative pain catastrophizing scale (PCS) scores with risk factors for severe pain postoperatively | 24 hrs postoperatively
  risk factors include: Age, gender, BMI, socio-economic condition, preoperative anxiety

CONTACTS AND LOCATIONS:
Locations (1):
- BP Koirala Institute of Health Sciences (BPKIHS), Dharān, Koshi, Nepal

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Subedi A, Pokharel K, Sah BP, Chaudhary P. Association of preoperative pain catastrophizing with postoperative pain after lower limb trauma surgery. J Psychosom Res. 2021 Oct;149:110575. doi: 10.1016/j.jpsychores.2021.110575. Epub 2021 Jul 24. PMID 34371257